CLINICAL TRIAL: NCT02259153
Title: A Randomized Study to Assess the Effect of Different Fat Enriched Meats on the Hepatic Cholesterol Synthesis
Brief Title: Effect of Different Fat Enriched Meats on the Hepatic Cholesterol Synthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Aragones de Ciencias de la Salud (Other Government)
Responsible Party: Principal Investigator, Fernando Civeira, Professor, Instituto Aragones de Ciencias de la Salud
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CEICA;PI13-00106
Record Dates: First submitted 2014-10-01; First posted 2014-10-08 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2014-10

CONDITIONS: Lipid Metabolism Disorders; Sterols; Diet, High-Fat; Cholesterol; Fatty Acids; Hyperlipidemias
Keywords: Lipids; Non Cholesterol Sterols; Oxysterols; Cholesterol Metabolism
MeSH Terms: conditions — Lipid Metabolism Disorders; Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Lean red meat diet (Active Comparator): Participants were given 350 g per day of lean red meat to incorporate to their usual diet for ten days.
  Interventions: Behavioral: Changes in cholesterol metabolism; Other: Lean red meat diet
- Fat red meat diet (Active Comparator): Participants were given 350 g per day of fat red meat to incorporate to their usual diet for ten days.
  Interventions: Behavioral: Changes in cholesterol metabolism; Other: Fat red meat diet

INTERVENTIONS:
Behavioral: Changes in cholesterol metabolism
Other: Lean red meat diet
  Arms: Lean red meat diet
Other: Fat red meat diet
  Arms: Fat red meat diet

SUMMARY:
The objective of the study is to assess the effect of two diets with different fat composition on cholesterol metabolism. The study was a randomized cross-over trial where volunteers follow two study periods with different types of meat (lean and fat red meat) separately by a ten days wash-out period. At the beginning of the study and after the study periods the following parameters are determined: anthropometric (weight, waist, circumference and body mass index), blood pressure, dietary (72-hours dietary registry) and exercise assessments and biochemical analysis (total cholesterol, triglycerides, HDL cholesterol, LDL cholesterol, apolipoprotein A1, apolipoprotein B, iron, transferring, ferritin, uric acid, glucose, HbA1c and insulin). Serum concentration of non cholesterol sterols (sitosterol, campesterol, stigmasterol, desmosterol and lanosterol) and oxysterols (24S-hydroxycholesterol, 27-hydroxycholesterol and 7α-hydroxycholestenone) were measured by High Performance Liquid Chromatography tandem Mass Spectrometry in these subjects throughout along the study in order to demonstrate the effect of different red meat on the hepatic metabolism of cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* Normolipemic healthy subjects defined by levels of LDL cholesterol and triglycerides below the 90th percentile adjusted for age and sex.
* Diet and stable lifestyle with controllable feeding.

Exclusion Criteria:

* Pregnancy or intention of pregnancy during the study.
* Lipid lowering drugs in the last 3 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-03; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Changes in lipid profile | Baseline and after 10 days of intervention
Changes in non cholesterol sterols and oxysterols serum concentrations | Baseline and after 10 days of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Civeira, MD, PhD, Principal Investigator — Unidad de Lípidos/ Laboratorio de Investigación Molecular; Hospital Universitario Miguel Servet; Instituto Aragonés de Ciencias de la Salud (Zaragoza, Spain); Lucía Baila-Rueda, MSc, Principal Investigator — Unidad de Lípidos/ Laboratorio de Investigación Molecular; Hospital Universitario Miguel Servet; Instituto Aragonés de Ciencias de la Salud (Zaragoza, Spain)

REFERENCES:
- [Derived] Baila-Rueda L, Mateo-Gallego R, Perez-Calahorra S, Lamiquiz-Moneo I, de Castro-Oros I, Cenarro A, Civeira F. Effect of different fat-enriched meats on non-cholesterol sterols and oxysterols as markers of cholesterol metabolism: Results of a randomized and cross-over clinical trial. Nutr Metab Cardiovasc Dis. 2015 Sep;25(9):853-859. doi: 10.1016/j.numecd.2015.06.008. Epub 2015 Jun 23. PMID 26232911